CLINICAL TRIAL: NCT03462004
Title: Phase 1 Evaluation of a Live-Attenuated Human Parainfluenza Virus Type 3 Vectored Vaccine Candidate Expressing Ebolavirus Zaire Glycoprotein as the Sole Envelope Glycoprotein
Brief Title: Evaluating the Live-Attenuated Human Parainfluenza Virus Type 3 Vectored Vaccine Candidate Expressing Ebolavirus Zaire Glycoprotein as the Sole Envelope Glycoprotein
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: On hold due to pandemic
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 324
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Ebola Virus Disease
Keywords: Healthy Volunteer
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: HPIV3/ΔHNF/EbovZ GP vaccine (Experimental): Participants will receive two doses of 10^6.0 PFU/mL of HPIV3/ΔHNF/EbovZ GP vaccine on Days 0 and 28 (+28).
  Interventions: Biological: HPIV3/ΔHNF/EbovZ GP vaccine
- Cohort 1: Placebo (Placebo Comparator): Participants will receive two doses of placebo on Days 0 and 28 (+28).
  Interventions: Biological: Placebo
- Cohort 2: HPIV3/ΔHNF/EbovZ GP vaccine (Experimental): Participants will receive two doses of 10^7.0 PFU/mL of HPIV3/ΔHNF/EbovZ GP vaccine on Days 0 and 28 (+28).
  Interventions: Biological: HPIV3/ΔHNF/EbovZ GP vaccine
- Cohort 2: Placebo (Placebo Comparator): Participants will receive two doses of placebo on Days 0 and 28 (+28).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: HPIV3/ΔHNF/EbovZ GP vaccine — Administered intranasally
  Arms: Cohort 1: HPIV3/ΔHNF/EbovZ GP vaccine; Cohort 2: HPIV3/ΔHNF/EbovZ GP vaccine
Biological: Placebo — Administered intranasally
  Arms: Cohort 1: Placebo; Cohort 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, infectivity, and immunogenicity of two doses of the HPIV3/ΔHNF/EbovZ GP vaccine candidate when administered intranasally in healthy adults.

DETAILED DESCRIPTION:
This study will evaluate the safety, infectivity, and immunogenicity of two doses of the HPIV3/ΔHNF/EbovZ GP vaccine candidate when administered intranasally in healthy adults.

Participants will be enrolled sequentially in two cohorts. Participants in Cohort 1 will be randomly assigned to receive two doses of either 10^6.0 PFU/mL of HPIV3/ΔHNF/EbovZ-GP vaccine or placebo. The first dose will be given on Day 0 and the second dose will be given 4-8 weeks later. Participants in Cohort 2 will be randomly assigned to receive two doses of either 10^7.0 PFU/mL of HPIV3/ΔHNF/EbovZ-GP vaccine or placebo on Days 0 and 28.

Participants will be admitted to the inpatient unit 2 days prior to receiving their first dose of the vaccine or placebo. While in the inpatient unit, study procedures will include physical examinations, nasal washes, and blood collection. Participants will be discharged from the inpatient unit on Day 8 or thereafter once two consecutive rRT-PCR assay results are below the pre-determined threshold. An additional study visit will occur on Day 14.

On Day 26 (+28), participants will be readmitted to the inpatient unit, and will receive their second dose of the vaccine or placebo on Day 28 (+28). Participants will undergo the same study procedures that occurred during the first inpatient stay, and will be discharged 7 days after the second dose, or once the subject is without respiratory symptoms and rRT-PCR assay is below the pre-determined threshold (around Day 35). Additional study visits will occur on Days 42 ± 3, 56 ± 5, 84 ± 5, 112 ± 7, 180 ± 14, 270 ± 14, and 360 ± 30.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant females between 18 and 50 years of age inclusive
* General good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator
* Agree to storage of blood specimens for future research
* Available for the duration of the trial
* Able to demonstrate understanding of key study concepts, study rationale, and study participation requirements by scoring greater than or equal to 70% on a written comprehension assessment in less than or equal to 3 attempts.
* Willingness to participate in the study as evidenced by signing the informed consent document
* Female subjects of childbearing potential must agree to have used effective birth control methods beginning at least one month prior to vaccination, and continuing with 'per label/fully effective use' for the chosen method for the duration of the study, from amongst these:

  * pharmacologic/hormonal contraceptives, including oral, parenteral, subcutaneous, and transcutaneous delivery;
  * condoms with spermicide;
  * diaphragm with spermicide;
  * intrauterine device;
  * absolute abstinence from heterosexual intercourse as a matter of normal preferred lifestyle;
  * or must be surgically sterile, or must be age 50 AND have had no menses at all for at least one full year.
  * All females must provide samples for urine and serum pregnancy testing prior to enrollment (immediately prior to each vaccination), as well as a statement of menstrual history and a summary of all potentially reproductive sexual activity for the month prior to each vaccination, and at each study contact throughout the study, and report if they may be pregnant immediately.
* Willingness to refrain from blood donation during the course of the study
* Willingness to refrain from receiving other vaccines or investigational products during the first 4 months of the study after enrollment
* Willingness to follow admission and isolation requirements for the indicated duration per protocol.

Exclusion Criteria:

* Pregnancy as determined by a positive human choriogonadotropin (ß-HCG) test or history of recent unprotected intercourse in a woman of reproductive capacity
* Currently breastfeeding
* Evidence of clinically significant neurological, cardiac, pulmonary, hepatic, rheumatological, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* History of intranasal pathology or evidence of structural abnormalities of the sinuses or nasal cavity upon examination
* Behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, affects the subject's ability to understand and cooperate with the study protocol
* Positive urine drug toxicology test indicating narcotic use or history of dependency
* Have medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial, or would render the subject unable to comply with the protocol.
* History of anaphylaxis
* Current diagnosis of asthma or reactive airway disease (within the past 2 years)
* Current history of allergic rhinitis requiring the use of medication in the 2 weeks before enrollment or the first 56 days of the study
* History of Bell's palsy
* Positive enzyme-linked immunosorbent assay (ELISA) and confirmatory test (e.g., Western blot or HIV-1/HIV-2 differentiation assay) for human immunodeficiency virus-1 (HIV-1)
* Positive ELISA and confirmatory test (e.g., polymerase chain reaction (PCR) for virus) for hepatitis C virus (HCV)
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA test
* Known immunodeficiency syndrome or history suggestive of impaired immune function
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination
* History of asplenia.
* Body mass index (BMI) less than 18.5 or greater than 40
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination
* Current tobacco user unwilling to refrain from smoking, snuffing, vaping, or chewing for the duration of the inpatient study (subjects may use nicotine patches if needed)
* Travel to an Ebola-endemic region at the time when cases were present or planned travel to West or Central Africa during the study period
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination
* Previous receipt of an investigational Ebola or Marburg virus vaccine, a chimpanzee adenovirus, or human parainfluenza virus (HPIV)-vectored vaccine, or any other investigational vaccine likely to affect interpretation of the trial data
* Current or past (in the last 4 weeks) user of intranasal medications (including steroids, decongestants, or hormonal medications), or planning to use them within 28 days of study vaccination
* Live or have close contact with vulnerable individuals, including infants, the elderly, or immunocompromised individuals (those with HIV/AIDS, malignancy, or transplant patients)
* History of Liver disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of vaccine-related solicited adverse events | Measured through Day 35
  Graded according to Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, March 2017
Area under the curve of nasal virus shedding after each dose of vaccine | Measured through Day 35
  Assessed by liquid titration of nasal secretions on LLC-MK2 monkey kidney cells
Development of serum antibody to the EbovZ GP | Measured through Day 360
  As measured by enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research, Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - CIR Inpatient Unit, Johns Hopkins Bayview Medical Center, Baltimore, Maryland

DOCUMENTS (1):
  • Informed Consent Form (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT03462004/ICF_000.pdf